CLINICAL TRIAL: NCT05372302
Title: Collecting Ducts Carcinoma: in Depth Exploration and Biologically Driven Therapy (CICERONE)
Acronym: CICERONE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Sponsor
Other Study IDs: INT 12/21
Record Dates: First submitted 2022-05-09; First posted 2022-05-12 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Collecting Duct Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
* Collect a large number of samples with certain / suspected diagnosis of collecting duct carcinoma in order to confirm the diagnosis (centralized review) and standardize according to WHO 2016 criteria
* Build an extensive tissue bank (DNA and RNA extraction) aimed at defining the molecular taxonomy of the tumor through 1) transcriptomic analysis 2) gene expression profile
* Define specific molecular signatures

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Signature of consent (for patients enrolled in the prospective part of the study)
* Histological diagnosis of renal cell carcinoma of the Bellini collecting duct RCC

Exclusion Criteria:

-

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with certain / suspected diagnosis of carcinoma of the collecting ducts
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-07-08 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
samples to confirm and standardize | 15 month
  Collect a large number of samples with certain / suspected diagnosis of collecting duct carcinoma in order to confirm the diagnosis (centralized review) and standardize it according to WHO 2016 criteria

SECONDARY OUTCOMES:
Tissue Bank | 15 month
  Build an extensive tissue bank (DNA and RNA extraction) aimed at defining the molecular taxonomy of the tumor through 1) transcriptomic analysis 2) gene expression profile
specific molecular signatures | 15 month
  Define specific molecular signatures

CONTACTS AND LOCATIONS:
Overall Officials: Filippo De Braud, Prof, Principal Investigator — Fondazione IRCCS Istituto Nazionale Tumori - Milano
Locations (1):
- Fondazione IRCCS Istituto Nazionale Tumori, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tokuda N, Naito S, Matsuzaki O, Nagashima Y, Ozono S, Igarashi T; Japanese Society of Renal Cancer. Collecting duct (Bellini duct) renal cell carcinoma: a nationwide survey in Japan. J Urol. 2006 Jul;176(1):40-3; discussion 43. doi: 10.1016/S0022-5347(06)00502-7. PMID 16753362
- [Background] Becker F, Junker K, Parr M, Hartmann A, Fussel S, Toma M, Grobholz R, Pflugmann T, Wullich B, Strauss A, Behnes CL, Otto W, Stockle M, Jung V. Collecting duct carcinomas represent a unique tumor entity based on genetic alterations. PLoS One. 2013 Oct 22;8(10):e78137. doi: 10.1371/journal.pone.0078137. eCollection 2013. PMID 24167600
- [Background] Gupta R, Billis A, Shah RB, Moch H, Osunkoya AO, Jochum W, Hes O, Bacchi CE, de Castro MG, Hansel DE, Zhou M, Vankalakunti M, Salles PG, Cabrera RA, Gown AM, Amin MB. Carcinoma of the collecting ducts of Bellini and renal medullary carcinoma: clinicopathologic analysis of 52 cases of rare aggressive subtypes of renal cell carcinoma with a focus on their interrelationship. Am J Surg Pathol. 2012 Sep;36(9):1265-78. doi: 10.1097/PAS.0b013e3182635954. PMID 22895263
- [Background] Selli C, Amorosi A, Vona G, Sestini R, Travaglini F, Bartoletti R, Orlando C. Retrospective evaluation of c-erbB-2 oncogene amplification using competitive PCR in collecting duct carcinoma of the kidney. J Urol. 1997 Jul;158(1):245-7. doi: 10.1097/00005392-199707000-00079. PMID 9186368
- [Background] Malouf GG, Comperat E, Yao H, Mouawad R, Lindner V, Rioux-Leclercq N, Verkarre V, Leroy X, Dainese L, Classe M, Descotes JL, Barthelemy P, Yacoub M, Roupret M, Bernhard JC, Creighton CJ, Spano JP, Su X, Khayat D. Unique Transcriptomic Profile of Collecting Duct Carcinomas Relative to Upper Tract Urothelial Carcinomas and other Kidney Carcinomas. Sci Rep. 2016 Aug 3;6:30988. doi: 10.1038/srep30988. PMID 27484008
- [Background] Wang J, Papanicolau-Sengos A, Chintala S, Wei L, Liu B, Hu Q, Miles KM, Conroy JM, Glenn ST, Costantini M, Magi-Galluzzi C, Signoretti S, Choueiri T, Gallucci M, Sentinelli S, Fazio VM, Poeta ML, Liu S, Morrison C, Pili R. Collecting duct carcinoma of the kidney is associated with CDKN2A deletion and SLC family gene up-regulation. Oncotarget. 2016 May 24;7(21):29901-15. doi: 10.18632/oncotarget.9093. PMID 27144525
- [Background] Pal SK, Choueiri TK, Wang K, Khaira D, Karam JA, Van Allen E, Palma NA, Stein MN, Johnson A, Squillace R, Elvin JA, Chmielecki J, Yelensky R, Yakirevich E, Lipson D, Lin DI, Miller VA, Stephens PJ, Ali SM, Ross JS. Characterization of Clinical Cases of Collecting Duct Carcinoma of the Kidney Assessed by Comprehensive Genomic Profiling. Eur Urol. 2016 Sep;70(3):516-21. doi: 10.1016/j.eururo.2015.06.019. Epub 2015 Jul 3. PMID 26149668
- [Background] Pagani F, Colecchia M, Sepe P, Apollonio G, Claps M, Verzoni E, de Braud F, Procopio G. Collecting ducts carcinoma: An orphan disease. Literature overview and future perspectives. Cancer Treat Rev. 2019 Sep;79:101891. doi: 10.1016/j.ctrv.2019.101891. Epub 2019 Aug 27. PMID 31491662
- [Background] Procopio G, Testa I, Iacovelli R, Grassi P, Verzoni E, Garanzini E, Colecchia M, Torelli T, De Braud F. Treatment of collecting duct carcinoma: current status and future perspectives. Anticancer Res. 2014 Feb;34(2):1027-30. PMID 24511050
- [Background] Procopio G, Verzoni E, Iacovelli R, Colecchia M, Torelli T, Mariani L. Is there a role for targeted therapies in the collecting ducts of Bellini carcinoma? Efficacy data from a retrospective analysis of 7 cases. Clin Exp Nephrol. 2012 Jun;16(3):464-7. doi: 10.1007/s10157-012-0589-3. Epub 2012 Jan 26. PMID 22278601
- [Background] G.Procopio, R. Ratta, G. Fucà, P. Grassi, L. Porcu, M. Prisciandaro, G. Calareso, R. Montone, M. Sorrentino, E. Verzoni. A phase 2 study of cabozantinib as first-line treatment in collecting ducts renal cell carcinoma: The BONSAI trial. J Clin Oncol 36, 2018.DOI:10.1200/JCO.2018.36.6_suppl.TPS709
- [Background] Liu L, Miao L, Liu Y, Qi A, Xie P, Chen J, Zhu H. S100A11 regulates renal carcinoma cell proliferation, invasion, and migration via the EGFR/Akt signaling pathway and E-cadherin. Tumour Biol. 2017 May;39(5):1010428317705337. doi: 10.1177/1010428317705337. PMID 28513300
- [Background] McDermott DF, Huseni MA, Atkins MB, Motzer RJ, Rini BI, Escudier B, Fong L, Joseph RW, Pal SK, Reeves JA, Sznol M, Hainsworth J, Rathmell WK, Stadler WM, Hutson T, Gore ME, Ravaud A, Bracarda S, Suarez C, Danielli R, Gruenwald V, Choueiri TK, Nickles D, Jhunjhunwala S, Piault-Louis E, Thobhani A, Qiu J, Chen DS, Hegde PS, Schiff C, Fine GD, Powles T. Clinical activity and molecular correlates of response to atezolizumab alone or in combination with bevacizumab versus sunitinib in renal cell carcinoma. Nat Med. 2018 Jun;24(6):749-757. doi: 10.1038/s41591-018-0053-3. Epub 2018 Jun 4. PMID 29867230
- [Background] Filipazzi P, Valenti R, Huber V, Pilla L, Canese P, Iero M, Castelli C, Mariani L, Parmiani G, Rivoltini L. Identification of a new subset of myeloid suppressor cells in peripheral blood of melanoma patients with modulation by a granulocyte-macrophage colony-stimulation factor-based antitumor vaccine. J Clin Oncol. 2007 Jun 20;25(18):2546-53. doi: 10.1200/JCO.2006.08.5829. PMID 17577033
- [Background] Huber V, Vallacchi V, Fleming V, Hu X, Cova A, Dugo M, Shahaj E, Sulsenti R, Vergani E, Filipazzi P, De Laurentiis A, Lalli L, Di Guardo L, Patuzzo R, Vergani B, Casiraghi E, Cossa M, Gualeni A, Bollati V, Arienti F, De Braud F, Mariani L, Villa A, Altevogt P, Umansky V, Rodolfo M, Rivoltini L. Tumor-derived microRNAs induce myeloid suppressor cells and predict immunotherapy resistance in melanoma. J Clin Invest. 2018 Dec 3;128(12):5505-5516. doi: 10.1172/JCI98060. Epub 2018 Nov 5. PMID 30260323
- [Background] E. Verzoni, S. Ferro, G. Procopio, A. Cova, R. Ratta, A. Raimondi, P. Sepe, P. Squarcina, L. Lalli, V. Huber, D. Rinchai, D. Bedognetti, L. Rivoltini. Potent Natural Killer (NK) and myeloid blood cell remodeling by Cabozantinib (Cabo) in pretreated metastatic renal cell carcinoma (mRCC) patients (pts). Annals of Oncology (2018) 29 (suppl_8): viii303-viii331.
- [Background] E. Verzoni, L. De Cecco, M. Dugo, D. Rinchai, D. Bedognetti, P. Grassi, R. Ratta, A. Cova, P. Squarcina, V. Huber, R. Montone, M. Sorrentino, G. Procopio, L. Rivoltini. Broad immunomodulating effect of first-line Pazopanib in metastatic renal cell carcinoma patients. Annals of Oncology (2017) 28 (suppl_5): v295-v329.
- [Background] Paquet ER, Hallett MT. Absolute assignment of breast cancer intrinsic molecular subtype. J Natl Cancer Inst. 2014 Dec 4;107(1):357. doi: 10.1093/jnci/dju357. Print 2015 Jan. PMID 25479802
- [Background] Cherkasova E, Scrivani C, Doh S, Weisman Q, Takahashi Y, Harashima N, Yokoyama H, Srinivasan R, Linehan WM, Lerman MI, Childs RW. Detection of an Immunogenic HERV-E Envelope with Selective Expression in Clear Cell Kidney Cancer. Cancer Res. 2016 Apr 15;76(8):2177-85. doi: 10.1158/0008-5472.CAN-15-3139. Epub 2016 Feb 9. PMID 26862115
- [Background] Dobin A, Davis CA, Schlesinger F, Drenkow J, Zaleski C, Jha S, Batut P, Chaisson M, Gingeras TR. STAR: ultrafast universal RNA-seq aligner. Bioinformatics. 2013 Jan 1;29(1):15-21. doi: 10.1093/bioinformatics/bts635. Epub 2012 Oct 25. PMID 23104886
- [Background] Procopio G, Sepe P, Claps M, Buti S, Colecchia M, Giannatempo P, Guadalupi V, Mariani L, Lalli L, Fuca G, de Braud F, Verzoni E. Cabozantinib as First-line Treatment in Patients With Metastatic Collecting Duct Renal Cell Carcinoma: Results of the BONSAI Trial for the Italian Network for Research in Urologic-Oncology (Meet-URO 2 Study). JAMA Oncol. 2022 Jun 1;8(6):910-913. doi: 10.1001/jamaoncol.2022.0238. PMID 35420628